CLINICAL TRIAL: NCT05146466
Title: Enhancing Men's Awareness of Testicular Diseases (E-MAT): A Feasibility Trial
Acronym: E-MAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Health Research Board, Ireland (Other); Health Research Board - Trials Methodology Research Network (Other)
Responsible Party: Principal Investigator, Mohamad Saab, Lecturer, University College Cork
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21125; DIFA-2020-028 (Other Grant/Funding Number: Health Research Board)
Record Dates: First submitted 2021-10-29; First posted 2021-12-06 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Testicular Diseases
Keywords: Testicular Diseases; Technology; Athletes; Knowledge; Social Media; Virtual Reality
MeSH Terms: conditions — Testicular Diseases

STUDY DESIGN:
Intervention Model Description: Data will be collected in up to 12 Gaelic Athletic Association (GAA) sports clubs. For each of the participating GAA clubs, individual participants will be randomised with the same probability to one of the two arms (E-MATVR [intervention]/E-MATE [control]). Allocation concealment will be maintained using a computerised system. Once participants have consented and their baseline assessment has been entered into the computer database, their allocation will be given by automated email. Randomisation and allocation concealment will be conducted according to the standard operating procedures (SOPs) of the Statistics and Data Analysis Unit of the HRB Clinical Research Facility-Cork (HRB CRF-C).
Masking Description: Given the differences between the two arms, participants will be aware of the arm they have been randomised into. Outcome assessments will be self-reported and returned to research staff with no information on allocation. Blinding will be maintained throughout data analysis. Unblinding will be facilitated by the independent statistician following completion of the protocol-specified data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-MATVR (intervention) (Other)
  Interventions: Behavioral: E-MATVR
- E-MATEE (control) (Other)
  Interventions: Behavioral: E-MATE

INTERVENTIONS:
Behavioral: E-MATVR — It involves using computer software uploaded onto wireless virtual reality (VR) technology (similar to downloading an app on a mobile phone) and will be delivered using a headset, handheld controllers, and voiceover (all wireless). E-MATVR comprises three serious gaming levels aimed at familiarising men with the normal look and feel of the testes, common testicular symptoms and diseases, and the importance of early help-seeking.
  Arms: E-MATVR (intervention)
Behavioral: E-MATE — It involves using the same information as EMATVR delivered as plain text (e.g., PDF) with still images from E-MATVR. Participants will be given approximately 10 minutes to read the text/look at images using a tablet (e.g., iPad).
  Arms: E-MATEE (control)

SUMMARY:
Hypothesis: Is it feasible to conduct a definitive trial to test the effect of E-MATVR compared to E-MATE on primary and secondary outcomes among Gaelic Athletic Association (GAA) members (players and coaches)?

The overall aim of this study is to examine the feasibility of conducting a definitive trial to test the effect of an educational intervention to Enhance Men's Awareness of Testicular diseases using Virtual Reality (E-MATVR) among male GAA members.

The effect of E-MATVR will be compared to E-MATE (control) which involves using the same information as E-MATVR delivered as plain text (e.g., PDF) with still images from E-MATVR.

DETAILED DESCRIPTION:
1. Overall aim

   To examine the feasibility of conducting a definitive trial to test the effect of E-MATVR (intervention) compared to Electronic information only, E-MATE (control) on testicular knowledge and testicular self-examination behaviours among male Gaelic Athletic Association (GAA) members (i.e., players and coaches) over three months.
2. Design

   According to Eldridge and colleagues, "feasibility study" is an umbrella term including randomised/non-randomised pilot studies and/or other feasibility studies aimed to determine whether a definitive trial can be done, should be done, and if so, how? To answer these questions, we the investigators will conduct a feasibility study comprising a feasibility trial, a study within a trial (SWAT), process evaluation and economic evaluation. This registration only contains the detailed description of the protocol for the feasibility trial.

   A Study Within A Trial (SWAT) will be conducted prior to the feasibility trial to determine which recruitment method (Twitter, Facebook or Quick Response [QR] code [via distributed leaflet]) is more efficient and cost effective for recruiting men to this feasibility study. A protocol for the SWAT is available in the SWAT Repository hosted at Queen's University Belfast (insert once available).

   A mixed- method process evaluation will be conducted to explore participants' experiences of E-MATVR and E-MATE and potential sources of intervention failure. A protocol for the process evaluation is available in HRB Open Research (insert once available)

   An economic evaluation will also be conducted to compare incremental costs and benefits of E-MATVR with E-MATE. A cost-benefit analysis will be employed whereby the costs and benefits will be measured in monetary terms. Data for the economic evaluation will be collected within the outcomes measures for the feasibility trial at T1 (immediately post-test) and T2 (three months follow up).
3. Objectives

   1. Negotiate access with key stakeholders.
   2. Identify unforeseen problems and safety issues.
   3. Examine randomisation and blinding processes.
   4. Provide estimates for sample size calculation for definitive trial.
4. Design

   Randomised feasibility trial.
5. Participants

   5.1 Inclusion criteria
   1. Biological males
   2. Members of the target GAA clubs since testicular injuries are common in field sports like hurling.
   3. Residing in Ireland.
   4. Aged 18-50 years (age group at risk for testicular diseases).

   5.2 Exclusion criteria
   1. History of seizures.
   2. History of motion sickness.
6. Setting

   Data will be collected in up to 12 geographically dispersed GAA clubs, including "Healthy Club" https://www.gaa.ie/my-gaa/community-and-health/healthy-club/).
7. Intervention

   Intervention described below using the template for intervention description and replication (TIDieR) checklist.

   7.1 Brief name

   E-MATVR.

   7.2 Why?

   Limitations from the investigators previous research were (i) the inclusion of men from one university; (ii) short follow-up time; (iii) lack of randomisation/control group; (iv) lack of an economic evaluation; and (v) lack of process evaluation. These will be addressed in this project.

   7.3 What?

   E-MATVR is a computer software uploaded onto VR technology and delivered using a headset, handheld controllers, and voiceover (all wireless). The voiceover script is based on evidence from the investigators prior research and the Preconscious Awareness to Action theoretical framework. The script's readability score (83.4 on the Flesch-Kincaid test) indicates its suitability for sixth Graders.

   E-MATVR comprises three gaming levels and takes approximately 10min to complete. The user is required to complete one area to move to the next area. E-MATVR begins with a popping series of words (like opening movie credits) as the voiceover reads them out. These include light-hearted synonyms for the testes (e.g., balls, nuts, gonads). The word "nuts" rather than "testes" is used to engage men with this intimate/sensitive topic.
   * Area 1 involves a 3D space with two walnuts. The user is asked by the voiceover to move around the walnuts using the controllers, while providing facts about the normal size and shape of the testes. Three changes (lump, swelling, and pain [represented as flashing light]) then appear consecutively. These are accompanied with a humorous emotional response from the voiceover. The user must find all three changes to move to the next level.
   * Area 2: A 3D model of a testis is used and the spermatic cord, epididymis, and tumour are represented. The user is loaded into Level 2 on top of the testis. During this level, the voiceover links symptoms experienced in Level 1 to testicular structures. The spermatic cord lights up to indicate testicular torsion and a purple lump appears, indicating a growth.
   * Area 3: Key messages are reiterated by the voiceover using three icons: (i) a snowflake to remind participants that their testes are unique and highlight the importance of knowing what is normal for them; (ii) an infographic with the method for testicular self-examination; and (iii) a red cross to prompt participants to seek help for abnormalities and seek immediate attention for severe testicular pain.

   7.4 Who provided?

   E-MATVR was developed by Mr Eoghan Cooke (Collaborator and Research Assistant) within an MSc in Interactive Media supervised by Mr David Murphy (Co-Applicant). A Research Assistant (Mr Billy O'Mahony) with interactive media expertise will test E-MATVR.

   7.5 How?

   E-MATVR is delivered using the latest VR technology (Oculus Quest 2 https://www.oculus.com/quest-2/) to give users a life-like experience, with imbedded headphones and controllers that provide vibrational (haptic) feedback based on participants' actions. The use of VR is explained, and participants are exposed to a brief demonstration to practice the use of the technology. Participants are then exposed to E-MATVR.

   7.6 Where?

   E-MATVR (wireless) will be tested in the target GAA clubs.

   7.7 When?

   Participants will complete E-MATVR once. E-MATVR takes approximately 10min to complete.

   7.8 How much?

   The number of VR users worldwide was 171 million in 2018, as compared to 200,000 in 2014. Worldwide spending on VR and augmented reality will grow between 2019-2023, achieving a Compound Annual Growth Rate of 77% and delivering a 294 billion USD boost to global Gross Domestic Product by supporting education and training. VR device ownership and purchase intent are highest among men aged 18-39yrs. The surge in VR use led to significant price drops. High-quality VR equipment is available for €138-€462 (https://www.oculus.com/compare/).

   7.9 Tailoring/Modifications

   Should a newer VR technology emerge, the E-MATVR software can be readily transferred in full onto it.

   7.10 How well?

   User-friendliness, acceptability, and effectiveness (one-group pre-post pilot) of E-MATVR were tested with 68 university students. Participants perceived E-MATVR as fun, innovative, informative, memorable, and user-friendly. E-MATVR was successful in increasing men's knowledge of testicular diseases, intentions to seek help for symptoms, and testicular self-examination behaviours.
8. Control

   E-MATE (E for Electronic information) will serve as the control arm. It involves using the same information as E-MATVR delivered as plain text (e.g., PDF) with still images from E-MATVR. Participants will be given 10min to read the text/look at images using an iPad.
9. Outcomes

   9.1 Primary outcomes
   1. Testicular knowledge (Dichotomous)
   2. Testicular self-examination behaviours (Dichotomous)

   9.2 Secondary outcomes
   1. Testicular awareness (Likert scale)
   2. Help-seeking intentions (Likert scale)
   3. Implementation intentions (Likert scale)
   4. Perceived risk of testicular disorders (Likert scale)

   Outcomes will be measured at baseline (T0), immediately post-test (T1), and three months post-test (T2) using the Castor EDC software (https://www.castoredc.com/).

   A Research Assistant and/or Research Support Officer will be present to ensure participant safety. There is no in-person follow-up. Participants will be contacted (phone call/text message/email) to ensure completion of outcome measurement at T2. Non-respondents and those who withdraw will be considered lost to follow-up. Retention is key to ensuring power and internal validity. This will be addressed in the SWAT described below.
10. Sample size

    Given that the goal of a feasibility trial is to identify problems that would impede the conduct of a larger, definitive efficacy trial, the investigators set the sample size at 59 based on advice from Viechtbauer et al. (2015) which is aimed at being able to detect failures in study processes that would occur just 5% of the time (with 95% confidence). Bearing in mind a potential attrition rate of 25%, 74 participants will be recruited.
11. Randomisation and allocation concealment

    For each of the participating GAA clubs, individual participants will be randomised with the same probability to one of the two arms (E-MATVR/E-MATE). Allocation concealment will be maintained using a computerised system. Once participants have consented and their baseline assessment has been entered into the computer database, their allocation will be given by automated email. Randomisation and allocation concealment will be conducted according to the standard operating procedures (SOPs) of the Statistics and Data Analysis Unit of the HRB Clinical Research Facility-Cork (HRB CRF-C).
12. Blinding

    Given the differences between the two arms, participants will be aware of the arm they have been randomised into. Outcome assessments will be self-reported and returned to research staff with no information on allocation. Blinding will be maintained throughout data analysis. Unblinding will be facilitated by the independent statistician following completion of the protocol-specified data analysis.
13. Data analysis

    Analyses will be conducted by the lead statistician, under the SOPs of the Statistics and Data Analysis Unit of the HRB CRF-C. Before recruitment, a detailed Statistical Analysis Plan will be uploaded alongside the study protocol to the relevant registries. Data will undergo extensive quality checking and potential errors will be verified from source data a priori.

    Analyses of outcomes will be conducted on an intention-to-treat basis. Differences in outcomes by study arm, over time, will be estimated using generalised linear mixed effects models with the appropriate link function (based on the distribution of the outcome or expected error distribution). The investigators will report minimally adjusted models, which will include effects of intervention arm and time. The investigators will report a fully adjusted model that includes the key predictor variables collected at baseline. Missing data will be evaluated and addressed using appropriate methods (e.g., multiple imputation or inverse-probability weighting). Effect estimates for all pre-specified primary and secondary endpoints, will be publicly reported with 95%CI and exact p-values, in accordance with recent guidance from the American Statistical Association.

    Analyses will be conducted using transparent, open-science tools. All analysis steps, including cleaning or modifications to study database, will be fully scripted and replicable. Scripts for the key analyses will undergo testing prior to data analysis. Upon completion, the study database will be prepared according to FAIR data principles and be made available along-side the analysis scripts.
14. Ethical considerations

This study will be conducted in line with ethical principles depicted in the Declaration of Helsinki. Ethical approval will be sought from the Clinical Research Ethics Committee at UCC. Participants will be provided with an information leaflet and will sign informed consent.

Participants will be asked to check with their General Practitioner for abnormalities (e.g., lump) identified during testicular self-examination. Participants will also be asked to visit the emergency department for sudden and severe testicular pain which is often associated with emergencies such as testicular torsion.

ELIGIBILITY:
Inclusion Criteria:

1. Biological males.
2. Members of the target GAA clubs (GAA players and coaches) since testicular injuries are common in field sports like hurling.
3. Residing in Ireland.
4. Aged 18-50 years (age group at risk for testicular diseases).

Exclusion Criteria:

1. History of seizures.
2. History of motion sickness.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The current project involves awareness of male-specific diseases (i.e. testicular diseases). Therefore, cis (biological) males, transwomen (male to female), and non-binary/gender nonconforming/gender neutral individuals who are biologically male will be eligible for inclusion. Individuals who are not biologically male will be welcome to interact with E-MATVR/E-MATE if desired; however, their participation will not be recorded.
Enrollment: 74 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Testicular Knowledge Questionnaire | T0 (baseline), T1 (immediately post-test), T2 (three months post-test)
  Change in participants' knowledge of the normal testes, testicular symptoms, testicular self-examination, and testicular diseases as assessed by the Testicular Knowledge Questionnaire comprising 8 multiple choice questions and 4 'True' and 'False' type questions. All 12 items are dichotomised into "Correct=1" and "Incorrect/Don't know=0." Scores range between 0 and 12. Higher scores indicate greater knowledge.
Testicular Self-Examination Behaviour Questionnaire | T0 (baseline), T2 (three months post-test)
  Change in participants' behaviours in relation to feeling their own testes and advising at least one man to do the same as assessed by the Testicular Self-Examination Behaviour Questionnaire comprising 3 'Yes' and 'No' type questions. All items are dichotomous: "Yes=1" and "No=0."

SECONDARY OUTCOMES:
Testicular Awareness Scale | T0 (baseline), T1 (immediately post-test), T2 (three months post-test)
  Change in participants' familiarity with their own testes, what normal and what is not normal, and ability to differentiate between what is normal and what is not normal as assessed by the 5-item Testicular Awareness Scale (5-point Likert scale). Scores range between 1 (Strongly Disagree) and 5 (Strongly Agree). Higher scores indicate greater testicular awareness.
Implementations Intentions Scale | T0 (baseline), T1 (immediately post-test), T2 (three months post-test)
  Change in participants' intentions to purposefully feel their own testes at least once over a one-month period and advising at least one man to do the same as assessed by the 3-item Implementations Intentions Scale (5-point Likert scale). Scores range between 1 (Strongly Disagree) and 5 (Strongly Agree). Higher scores indicate greater implementation intentions.
Perceived Risk Item | T0 (baseline), T1 (immediately post-test), T2 (three months post-test)
  Change in participants' perceived risk of developing a testicular disease as assessed by the Perceived Risk Item (5-point Likert scale). Scores range between 1 (Strongly Disagree) and 5 (Strongly Agree). Higher scores indicate greater perceived risk.
General Help-Seeking Questionnaire | T0 (baseline), T1 (immediately post-test), T2 (three months post-test)
  Change in participants intentions to seek help for three testicular symptoms from different sources as assessed by the 3-item General Help-Seeking Questionnaire (7-point Likert scale). Scores range between 1 (Extremely Unlikely) and 7 (Extremely Likely) for each symptom. Higher scores indicate greater intentions to seek help.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad M Saab, PhD, MSc, PGDTLHE, RGN, Principal Investigator — University College Cork
Locations (1):
- Up to 12 geographically dispersed GAA clubs in Cork and neighbouring counties, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089
- [Derived] Murphy A, Kirby A, De Blasio F, McCarthy M, Shiely F, Hegarty J, Davoren MP, Harrington JM, Shorter GW, Murphy D, O'Mahony B, Cooke E, Rovito MJ, Robertson S, FitzGerald S, Connor AO, Riordan MO, Saab MM. Cost-Benefit Analysis of the Enhancing Men's Awareness of Testicular diseases (E-MAT) Feasibility Trial: A Virtual Reality Experience to Increase Testicular Knowledge and Self-Examination among Male Athletes. Pharmacoecon Open. 2025 Jul;9(4):671-682. doi: 10.1007/s41669-025-00571-5. Epub 2025 Mar 19. PMID 40108097
- [Derived] Saab MM, McCarthy M, Davoren MP, Shiely F, Harrington JM, Shorter GW, Murphy D, O'Mahony B, Cooke E, Murphy A, Kirby A, Rovito MJ, Robertson S, FitzGerald S, O'Connor A, O'Riordan M, Hegarty J, Dahly D. Enhancing Men's Awareness of Testicular Diseases (E-MAT) using virtual reality: A randomised pilot feasibility study and mixed method process evaluation. PLoS One. 2024 Jul 22;19(7):e0307426. doi: 10.1371/journal.pone.0307426. eCollection 2024. PMID 39037976
- See also: Related Info — https://www.gaa.ie/my-gaa/community-and-health/healthy-club/.
- See also: Related Info — https://www.oculus.com/quest-2.
- See also: Related Info — https://www.oculus.com/compare/